CLINICAL TRIAL: NCT03783832
Title: Follow up of Diabetic Macular Edema Treated by Aflibercept (Eylea®) With OCT-Angiography
Acronym: DOCTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aquitania Opthalmologica (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A03478-45
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: OCT ANGIOGRAPHY DATA — Follow-up of diabetic macular edema treated by Aflibercept (EYLEA®) with OCT angiography

SUMMARY:
This is a non-interventional, longitudinal, retrospective and prospective, non-controlled, single arm study in naive or non-naive patients with diabetic macular edema for which aflibercept (EYLEA®) therapy is indicated.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 years and more under reliable method of contraception for woman with childbearing potential (hormonal or any intrauterine devices).
* Patients with type I or II diabetes (as defined by criteria of American diabetes association ADA or world health organization WHO) with an glycosylated hemoglobin rate (HbA1c) < 10.0%, at initial visit (First EYLEA® injection).
* Patients with diabetes treatment unchanged within the last 3 months prior to initial visit (First EYLEA® injection).
* Patients showing a visual lost due to a diabetic macular edema (DME) in the central region and not for another reason, assessed by the investigateur. The visual acuity of the fellow eye is not an exclusion criteria.
* Patient to whom a treatment by aflibercept is indicated and OCT-angiography is performed at each injection visit.
* Patients affiliated to social security system.
* Patient who has been given appropriate information about the study objectives and instructions who has given his/her non-opposition prior to conduct any study-related procedures and examination.

Non iclusion Criteria:

* Treatment with an anti VEGF (EYLEA®, LUCENTIS® or AVASTIN®) administrated by intravitreal injection within 3 months prior to initial visit in the study eye
* Treatment with Ozurdex® administrated by intravitreal injection within 6 months prior to initial visit (First EYLEA® injection) in the study eye
* History of or active ocular /intraocular inflammation (Uveitis) at initial visit (First EYLEA® injection), in either eye
* Intra-ocular pressure ≥ 25 mmHg
* Patient with neocascular glaucoma history
* Patient with foveolar exsudat that interfere with images analysis.
* History or current evidence of hypersentivity to mydriatic eye drops
* Vitreomacular traction in the study eye
* Panretinal coagulation within 3 months prior to initial visit (First EYLEA® injection), in the study eye.
* Cataract surgery in the study eye within the 6 months prior to initial visit (First EYLEA® injection)
* History of vitretectomy in the study eye
* Treatment with systemic anti VEGF medications for cancer
* History of cerebrovascular accident within 3 months prior to initial visit (First EYLEA® injection), renal failure, uncontrolled arterial hypertension (PAS>160 mm Hg and/ or PAD>100 mm Hg)
* Patient who does not meet the local indication criteria for Eylea® treatment. Contraindications listed in the SmPCs must be taken into account
* Participation in any investigational study with exclusion period in progress at the initial visit (First EYLEA® injection)
* Patients under guardianship
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Diabetic Macular Edema
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative data from OCT angiography | 1 Year
  The macular perfusion measurement with Foveal Avascular Zone assessment (area in mm2, boundary in mm, circularity in %) measured by OCT angiography
Quantitative data from OCT angiography | 1 Year
  The perfusion density assessment (%) measured by OCT angiography
Quantitative data from OCT angiography | 1 Year
  The vascular density assessment (%) measured by OCT angiography

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU Bordeaux, Bordeaux
  - CHU Dijon, Dijon
  - Hôpital de la Croix-Rousse, Lyon
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - CHU Strasbourg, Strasbourg